CLINICAL TRIAL: NCT06491433
Title: A Prospective, Single Arm, Single Center, Non-randomized, Open Label Study to Evaluate the Accuracy of the Wrist Blood Pressure Monitor (H2-BP) Comparing With Aneroid Sphygmomanometer
Brief Title: Clinical Trial of H2-BP Electronic Sphygmomanometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Byoung Kwon Lee, Professor, Gangnam Severance Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2022-0427
Record Dates: First submitted 2024-06-30; First posted 2024-07-09 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Low Blood Pressure; Normal Blood Pressure; Prehypertension; Hypertension
MeSH Terms: conditions — Hypotension; Prehypertension; Hypertension | interventions — Sphygmomanometers; Blood Pressure Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test subjects using H2-BP and big ben® Sphygmomanometer (Experimental): Blood Pressure Measurement with the H2-BP Electronic Sphygmomanometer (H2-BP) and with aneroid Sphygmomanometer(big ben® Sphygmomanometer).
  Interventions: Device: H2-BP

INTERVENTIONS:
Device: H2-BP — The patient will have the test device applied to one wrist to measure blood pressure and the control device applied to the upper arm of the same arm to measure blood pressure.
  1. H2-BP: The test device is placed on the wrist and presses a button to start pressurising. When the measurement is complete, the systolic and diastolic blood pressure is displayed on the screen.
  2. big ben® Sphygmomanometer: The cuff is placed on the upper arm and the pump is pressed manually to inflate. 2 measurers will measure systolic and diastolic blood pressure by connecting 2 stethoscopes separately to one cuff.
  Due to the external nature of the study medical device, it is not possible to blind subjects and investigators, so that subjects and measurers are aware of the allocation. Therefore, blinding of subjects and measurers will not be used in this study.
  Other Names: Sphygmomanometer; Blood Pressure Measurement

SUMMARY:
The study compares H2-BP, a wristband blood pressure monitor, with an auscultatory sphygmomanometer. Both devices are used on the same arm. After confirming wrist and upper arm circumference, H2-BP is operated by one measurer, while the auscultatory sphygmomanometer is simultaneously operated by two other measurers. Each subject undergoes alternating measurements of H2-BP on one wrist and the auscultatory sphygmomanometer on the same arm until three valid measurement pairs are obtained per subject, with a maximum of eight repetitions allowed. The two auscultatory sphygmomanometer measurers operate independently and cannot see each other's measurements during the test. Measurements are repeated for 10 to 30 minutes until three valid blood pressure values are obtained and recorded. Validity assessment variables are derived from the recorded values to evaluate the accuracy of H2-BP.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients and inpatients aged 19 years or older showing hypotension, normal blood pressure, prehypertension, and hypertension
* Individuals who meet the criteria for wrist circumference, age, gender, and upper arm circumference as specified in the target number of participants.
* Those who have listened to a detailed explanation of the clinical trial, fully understand it, voluntarily decide to participate, and provide written consent to comply with precautions.

Exclusion Criteria:

* Patients who do not consent to participate in the study.
* Individuals who may not maintain stable blood pressure for approximately 30 minutes due to conditions resembling hypovolemia or similar conditions.
* Those who may not maintain stable blood pressure for approximately 30 minutes due to short-acting vasodilators or similar medications.
* Individuals with arrhythmia.
* Those who have eaten within 30 minutes before blood pressure measurement.
* Individuals who have consumed caffeine-containing beverages within 1 hour or smoked within 15 minutes before measurement.
* Participants who have exercised immediately before blood pressure measurement.
* Other patients deemed unsuitable for the study at the discretion of the researchers.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender Eligibility Description: At least 30% of the total participants must be composed of each gender (male and female)
Enrollment: 141 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital,, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Subjects Using H2-BP and Big Ben® Sphygmomanometer: Blood Pressure Measurement with the H2-BP Electronic Sphygmomanometer (H2-BP) and with aneroid Sphygmomanometer(big ben® Sphygmomanometer).
  H2-BP: The patient will have the test device applied to one wrist to measure blood pressure and the control device applied to the upper arm of the same arm to measure blood pressure.
  1. H2-BP: The test device is placed on the wrist and presses a button to start pressurising. When the measurement is complete, the systolic and diastolic blood pressure is displayed on the screen.
  2. big ben® Sphygmomanometer: The cuff is placed on the upper arm and the pump is pressed manually to inflate. 2 measurers will measure systolic and diastolic blood pressure by connecting 2 stethoscopes separately to one cuff.
  Due to the external nature of the study medical device, it is not possible to blind subjects and investigators, so that subjects and measurers are aware of the allocation. Therefore, blinding of subjects and measurers will not be used in this study.
Period: Overall Study
Arm/Group | Test Subjects Using H2-BP and Big Ben® Sphygmomanometer
Started | 141
Completed | 87
Not Completed | 54
Not completed — Protocol Violation | 51
Not completed — consent withdrawal | 2
Not completed — screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Test Subjects Using H2-BP and Big Ben® Sphygmomanometer
Number analyzed (Participants) | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 83
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.69 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 87
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean and Standard Deviation of Differences Between H2-BP Device and Aneroid Sphygmomanometer Measurements.
Description: Average difference between blood pressure measurements obtained with the test medical device and the comparator.
  Standard deviation of the difference between blood pressure measurements obtained with the test medical device and the comparator (based on the number of measurements).
Time Frame: serial assessment during 1 day
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Test Subjects Using H2-BP and Big Ben® Sphygmomanometer
Number analyzed (Participants) | 87
kPa
  systolic blood pressure | 0,276 (0,937)
  diastolic blood pressure | -0,004 (0,904)

2. Secondary Outcome: Standard Deviation of Differences Between H2-BP Device and Aneroid Sphygmomanometer Measurements.
Description: Standard deviation of the difference in blood pressure measurements between the test device and the comparator (based on the number of participants)
Time Frame: secondary outcome will be out in 1 day
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Test Subjects Using H2-BP and Big Ben® Sphygmomanometer
Number analyzed (Participants) | 87
kPa
  systolic blood pressure | 0,276 (0,789)
  diastolic blood pressure | -0,004 (0,735)

ADVERSE EVENTS:
Time Frame: 1day
Description: Death, serious adverse events, and other(non-serious adverse events) were not assessed for the study.
Arm/Group | Test Subjects Using H2-BP and Big Ben® Sphygmomanometer
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT06491433/Prot_SAP_000.pdf